CLINICAL TRIAL: NCT07306299
Title: An Exploratory Phase I Clinical Trial of a Universal mRNA Vaccine for Recurrent or Progressive High-grade Glioma
Brief Title: A Phase I Clinical Trial of a mRNA Vaccine for Recurrent or Progressive High-grade Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025LSYD1864
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Glioma, High Grade
Keywords: Glioma; mRNA vaccine; Mutation
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mRNA vaccine treatment group (Experimental): Participants in this arm receive the glioma-related multi-trageted mRNA vaccine.
  Interventions: Biological: Glioma-related multi-target mRNA vaccines

INTERVENTIONS:
Biological: Glioma-related multi-target mRNA vaccines — Multi-targeted mRNA vaccines encoding the following GBM-associated mutations: H3.3K27M, H3.1K27M, H3.3G34R, BRAFV600E, PIK3CAH1047R, IDH1R132H, EGFRvIII
  Other Names: mV002

SUMMARY:
This clinical trial is designed to evaluate the safety and efficacy of a universal mRNA vaccine targeting a panel of glioma-associated mutations in patients with recurrent or progressive high-grade glioma.

The primary objectives are to address the following key questions: 1) Is the mRNA vaccine safe for this patient population? 2) Does the vaccine stimulate an anti-tumor immune response and promote tumor regression?

Participants will receive the vaccine according to the following schedule:

1. one injection per week for four consecutive weeks, followed by one injection every four weeks for four cycles, and subsequently, one injection every 12 weeks for maintenance.
2. Safety and efficacy assessments, including detailed recording of adverse events and tumor growth evaluation, will be conducted at follow-up visits scheduled for weeks 6, 12, and months 6, 9, 12, 18, 24, and 36 post-treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate compliance, ability to comprehend the clinical trial, and provision of written informed consent.
2. Male or female, aged ≥16 years.
3. Histologically or cytologically confirmed WHO Grade III or IV glioma harboring one or more of the following mutations: H3.3K27M, H3.1K27M, H3.3G34R, BRAF V600E, PIK3CA H1047R, IDH1 R132H, or EGFRvIII.
4. Recurrent or progressive high-grade glioma, defined as a CNS WHO Grade 3-4 glioma confirmed by post-surgical histopathology, with documented recurrence or progression per RANO criteria on MRI following standard therapy (radiotherapy plus temozolomide chemotherapy).
5. Life expectancy ≥3 months.
6. Karnofsky Performance Status (KPS) ≥50. For subjects with spinal cord lesions, functional deficits due to paralysis will not be considered in the KPS assessment.
7. Absence of significant bone marrow, cardiac, pulmonary, or renal dysfunction, defined as:

   1. Hematologic (without transfusion or hematopoietic growth factor support within 14 days):

      * Absolute Neutrophil Count (ANC) ≥1.5 × 10⁹/L
      * Platelet count (PLT) ≥100 × 10⁹/L
      * Hemoglobin (HGB) ≥90 g/L
   2. Hepatic Function:

      * Alanine Aminotransferase (ALT) ≤2.5 × Upper Limit of Normal (ULN)
      * Aspartate Aminotransferase (AST) ≤2.5 × ULN
      * Total Bilirubin (TBIL) ≤1.5 × ULN
   3. Renal Function:

      * Serum creatinine ≤1.5 × ULN OR estimated creatinine clearance ≥50 mL/min (calculated using the Cockcroft-Gault formula)
   4. Coagulation:

      * Activated Partial Thromboplastin Time (APTT) ≤1.5 × ULN
      * International Normalized Ratio (INR) ≤1.5 × ULN
   5. Other:

      * Left Ventricular Ejection Fraction (LVEF) ≥50% without clinically significant pericardial effusion on echocardiogram
      * No clinically significant electrocardiogram (ECG) abnormalities
      * Baseline oxygen saturation >92% on room air
8. Adequate immune function, defined as receiving dexamethasone ≤2 mg/day within the 3 days prior to screening without severe lymphopenia.
9. Negative pregnancy test for women of childbearing potential (WOCBP); non-pregnant and non-lactating females; both male and female participants must agree to use highly effective contraception and have no plan for pregnancy within 6 months after study entry.

Exclusion Criteria:

1. History of other malignancies within the past 5 years (except appropriately treated carcinoma in situ of the cervix or non-melanoma skin cancer).
2. History of hypersensitivity to chemotherapy agents or radiosensitizers used for central nervous system or head and neck cancers.
3. History of severe allergic reactions to vaccines or any components of the investigational product.
4. Positive serology for:

   * Human Immunodeficiency Virus (HIV) antibody
   * Hepatitis C Virus (HCV) antibody with detectable HCV RNA
   * Hepatitis B Surface Antigen (HBsAg) with HBV DNA ≥2000 IU/mL
   * Treponema pallidum (TP) antibody with a positive confirmatory test (e.g., RPR/TPPA)
5. Active, uncontrolled infection, active tuberculosis, or active immunosuppressive disease.
6. Any concurrent non-malignant illness or psychiatric condition that would preclude safe protocol participation; uncontrolled cardiovascular disease (e.g., coronary artery disease, angina, myocardial infarction, significant arrhythmias).
7. Inability or unwillingness to provide informed consent or participate voluntarily.
8. Concurrent participation in another interventional clinical trial or participation within 3 months prior to screening.
9. Severe infection or signs/symptoms of active infection within 2 weeks prior to the first dose of the investigational product.
10. Administration of a live-attenuated vaccine within 4 weeks prior to the first dose.
11. History of solid organ or hematopoietic stem cell transplantation.
12. Any other condition that, in the opinion of the investigator, would jeopardize the subject's safety or compliance with the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a mRNA vaccine | 2-3 years
  All adverse events (AEs) treatment, emergent adverse events, treatment related toxici will be recorded. AE severity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version [Specify Version, e.g., 5.0]. Dose-limiting toxicities (DLTs) are defined as occurring within the DLT observation period [Specify period, e.g., 28 days after the first dose] and include:
  1. Any CTCAE Grade 4 local injection site reaction.
  2. Any CTCAE Grade 3 local injection site reaction persisting for ≥2 weeks despite optimal supportive care.
  3. Any hypersensitivity reaction of at least CTCAE Grade 3 severity.
  4. CTCAE Grade 4 cerebral edema.
  5. Autoimmune reactions of CTCAE Grade 3 or higher.
  6. Any CTCAE Grade 4 hematologic toxicity (e.g., neutropenia, thrombocytopenia, anemia).
  7. CTCAE Grade 3 or higher non-hematologic organ toxicity, with the following

SECONDARY OUTCOMES:
Immune response to mRNA vaccine | 1-5 years
  The proportion of activated T cells and IFN-γ content in the peripheral blood, and the T cell receptor (TCR) targeting each mutation were measured after mRNA vaccine treatment.

OTHER OUTCOMES:
Response rate to mRNA vaccine | 2-5 years
  The rates of OS and PFS assessed every 2 months until the end of the study. According to RECIST 1.1 criteria, the patients were divided into complete response (CR), partial response (PR), no change (SD: neither disease progression nor partial response compared with the sum of the minimum long diameters recorded since the beginning of treatment) and progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Zhu, M.D., Ph.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Room 521, Building 12, Jiefang Road Campus, The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: All